CLINICAL TRIAL: NCT01806285
Title: Sample Collection to Evaluate an Investigational Instrument for the Detection of Respiratory Viruses in Nasopharyngeal Swabs
Status: Completed | Type: Observational
Sponsor: GenMark Diagnostics (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP0001
Record Dates: First submitted 2013-02-26; First posted 2013-03-07 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Viral Respiratory Infection
Keywords: Respiratory Virus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Respiratory Symptoms

SUMMARY:
The purpose of this sample collection study is to prospectively collect respiratory viral clinical samples, conduct standard of care comparator testing and archive the collected residual samples for future testing in order to establish the clinical performance characteristics of the investigational instrument.

ELIGIBILITY:
Inclusion Criteria:

* The specimen is a nasopharyngeal swab.
* The specimen is from a pediatric or adult male or female subject who is either hospitalized, admitted to a hospital emergency department, visiting an outpatient clinic or resident of a long term care facility.
* The specimen is from a patient exhibiting clinical signs and symptoms of respiratory tract infection such as fever, sore throat, shortness of breath, bronchitis, bronchiolitis, and pneumonia.

Exclusion Criteria:

* The specimen is not a nasopharyngeal swab.
* The specimen is from an individual who does not exhibit clinical signs and symptoms of respiratory tract infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adults of any age suspected of having respiratory infection with onset of symptoms and fever within 5 days of sample collection.
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Sample collection study only | prospective sample collection